CLINICAL TRIAL: NCT03040895
Title: Effect Evaluation of The International Child Development Programme (ICDP)
Acronym: ICDP RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: Norwegian Directorate for Children, Youth and Family Affairs (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Public 360-nr. 16/13557
Record Dates: First submitted 2017-01-30; First posted 2017-02-02 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Parenting; Parent-Child Relations; Child Development
Keywords: Parenting practices
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICDP-intervention for caregivers (Experimental): Group-based ICDP-intervention for caregivers through a sequence of eight meetings. The groups are led by facilitators trained in the ICDP.
  Interventions: Other: Group-based ICDP-intervention
- Treatment as usual (Other): Participants may use other health services (GP, other interventions) as usual through the data Collection period (6 months). Afther this period, they will have the opportunity to join an ICDP-Group if they still want.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Group-based ICDP-intervention — Group-based ICDP-intervention for caregivers through a sequence of eight meetings
  Arms: ICDP-intervention for caregivers
Other: Treatment as usual — Treatment as usual through the data collection period (6 months)
  Arms: Treatment as usual

SUMMARY:
This study evaluate if a parental guidance programme based on the International Child Development Programme (ICDP) offered to the general Norwegian population, has an effect on caregivers, the relationship between caregiver and child, and on children's Development.

DETAILED DESCRIPTION:
The International Child Development Programme (ICDP) is a psychosocial preventive programme offered to parents and other caregivers. The programme aims to improve parenting practices and thereby child development and well-being. The ICDP is designed to influence and improve the quality of contact and relation between the caregivers, usually parents, and their children through the practical application of eight themes or guidelines for positive interaction. ICDP courses are implemented in a group format and include group discussions, caregiver assignments, and report back through a sequence of eight meetings. The caregiver groups are led by facilitators trained in the ICDP, and with the competence to lead such groups.

The aim of this study is to evaluate if ICDP has an effect on caregiver's positive involvement and sensitivity to childrens emotions, and on parental self-efficacy. The study will also evaluate the effect of ICDP on caregiver-child relationships, and the children's development and well-being.

The study will use a stratified cluster randomized control design, and will be implemented in regular clinical practice in Norway.

More knowledge within this field is important for practitioners as well as policy makers in planning preventive interventions for caregivers ant their children.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers with children between the age of 0-18 years, from the general Norwegian population
* Participants must be able to speak and write adequately Norwegian

Exclusion Criteria:

* Not having children between 0-18 years
* Insufficient Norwegian language skills
* ICDP imposed by resolution in the Fylkesnemnda

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 666 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Change in parents' reactions to children's emotions. Measurement: Coping With Toddlers'/Children's Negative Emotions Scale (CTNES/CCNES) | Assessment points: Baseline (just before the intervention), 10-12 weeks after baseline (immediately after the intervention), and 6 months after baseline
Change in positive Involvement with children. Measurement used: Alabama Parenting Questionnaire (APQ) | Assessment points: Baseline (just before the intervention), 10-12 weeks after baseline (immediately after the intervention), and 6 months after baseline
Change in Parenting self-efficacy. Measurement: Tool to measure Parenting Self Efficacy (TOPSE) | Assessment points: Baseline (just before the intervention), 10-12 weeks after baseline (immediately after the intervention), and 6 months after baseline

SECONDARY OUTCOMES:
Change in inter-parental conflict over child rearing issues. Measurement: Parenting Problem Checklist (PPC) | Assessment points: Baseline (just before the intervention), 10-12 weeks after baseline (immediately after the intervention), and 6 months after baseline
Change in the parent- child relationship. Measurement: Child-parent relationship scale (CPRS) | Assessment points: Baseline (just before the intervention), 10-12 weeks after baseline (immediately after the intervention), and 6 months after baseline
  Closeness and conflicts
Change in the child's psychosocial functioning. Measurement:Strength and Difficulties Questionnaire (SDQ) | Assessment points: Baseline (just before the intervention), 10-12 weeks after baseline (immediately after the intervention), and 6 months after baseline
  Emotional symptoms, hyperactivity, conduct problems, peer problems, prosocial behavior
Change in the child's quality of life. Measurement: KINDer und Jugendliche zur Erfassung der gesundheitsbezogenen Lebensqualität (KINDL) | Assessment points: Baseline (just before the intervention), 10-12 weeks after baseline (immediately after the intervention), and 6 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gun-Mette B. Røsand, PhD, Principal Investigator — Norwegian Institute of Public Health
Locations (1):
- Norwegian Institute of Public Health, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No